CLINICAL TRIAL: NCT07347652
Title: Development of a Nursing Care Protocol for the Prevention of Deep Vein Thrombosis and Its Impact on Patient Outcomes Following Cardiac Surgery
Brief Title: This Research Proposal Focuses on Evaluating the Effectiveness of a Nursing Care Protocol in Preventing Deep Vein Thrombosis (DVT) in Patients Undergoing On-pump Cardiac Surgery. The Study Will Include an Intervention Group That Receives the Nursing Protocol and a Control Group That Receives Routine
Acronym: DVT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Collaborators: Al-Ahli Hospital, Hebron (Unknown)
Responsible Party: Principal Investigator, Abdallah Ibraheem Abdallah Halahla, Development of a Nursing Care Protocol for the Prevention of Deep Vein Thrombosis and Its Impact on Patient Outcomes Following Cardiac Surgery, Near East University, Turkey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NEU\2025\138-2044
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: On-pump Cardiac Surgery - Prevention - Intervention - Experimental Group - Control Group - Incidence - Complications; DVT - Deep Vein Thrombosis; DVT Prophylaxis; DVT Prevention; Cardiac On-pump Surgery; Nursing Care Protocol
Keywords: DVT; NCP; CPS
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Experimental Group,Justification: The experimental group will receive a specific intervention aimed at preventing deep vein thrombosis (DVT) in on-pump cardiac surgery patients.
  * Sample Selection: Participants will be selected from a specific hospital or clinical setting based on predetermined inclusion and exclusion criteria.
  * Source of Sample: Patients admitted to the participating hospital or clinical setting for on-pump cardiac surgery.Control Group,Justification: The control group will serve as a comparison to evaluate the effectiveness of the intervention by comparing the occurrence of DVT in this group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing Care Protocol The nursing care protocol designed for this study is a structured, evidence-ba (Experimental): Nursing Care Protocol The nursing care protocol designed for this study is a structured, evidence-based guideline specifically tailored for on-pump cardiac surgery patients. It differs from existing DVT prevention protocols by integrating four core components: individualized risk stratification (using Padua and Caprini scores), combined pharmacological and mechanical prophylaxis, an early mobilization regimen adapted to post-cardiac surgery tolerance, and a structured patient education component. Unlike generic thromboprophylaxis guidelines, this protocol standardizes nursing-led interventions and monitoring across preoperative, intraoperative, and postoperative stages.
  Follow-Up Schedule and Time-Points
  Follow-Up Time-Points:
  * Day 0 (Start of prophylaxis / Baseline)
  * Day 3 (Early in-hospital monitoring)
  * Day 7 (or just before discharge)
  * Week 2 (Outpatient follow-up)
  * Month 3 (Long-term follow-up)
  Interventions: Device: IPC devices facilitate venous return by simulating the physiological effects of muscle contraction, reducing venous stasis.

INTERVENTIONS:
Device: IPC devices facilitate venous return by simulating the physiological effects of muscle contraction, reducing venous stasis. — Padua Prediction Score is a clinical tool that has been validated and created to identify hospitalized medical patients who are at risk of developing Venous Thromboembolism (VTE).
  Caprini's Risk Assessment Model (RAM) is one of the preferred risk scoring systems for assessing VTE chances for surgery patients. Joseph A. Caprini introduced it, which combines the hereditary and environmental risk factors, with a total of more than 40 different variables used in the assessment such as age, body mass index, past occurrence of VTE, varicose veins, presence of cancer, hormone therapy, and the length of immobility. The resulting score then puts patients into risk categories of very low with 0 points, low with 1-2 points, moderate with 3-4 pts., and high with ≥5 points.
  Other Names: Anticoagulant therapy reduces the likelihood of clot formation in high-risk individuals by inhibiting thrombus development.; Early identification of at-risk patients enables proactive preventive strategies, reducing the likelihood of complications.; Ambulation stimulates circulation and prevents venous stasis, a primary risk factor for DVT.; Proper hydration reduces blood viscosity, which helps prevent thrombosis.; Awareness empowers patients to recognize early warning signs and seek medical attention promptly.; Accurate record-keeping ensures continuity of care and facilitates early identification of potential complications.

SUMMARY:
The primary focus of this research proposal is to examine the efficacy of a nursing care protocol in preventing the occurrence of deep vein thrombosis (DVT) in patients undergoing on-pump cardiac surgery. The investigation will encompass an experimental group that will be subjected to a specific intervention, alongside a control group that will adhere to conventional care procedures. The central objective is to exhibit a statistically significant decrease in the incidence of DVT within the experimental group in comparison to the control group. The secondary outcomes involve assessing the severity of DVT instances and the development of associated complications.

The proposed research strategy entails delineating the criteria for selecting participants, outlining methodologies for gathering data, and detailing statistical approaches for analysis. The amassed data will undergo scrutiny through suitable statistical examinations, including chi-square tests, t-tests, or Mann-Whitney U tests, as well as logistic regression analysis. The process of data analysis will involve descriptive statistics, comparative assessments, regression analysis, and subgroup scrutiny. The interpretation of outcomes will be contextualized within the framework of the research objectives and pre-existing scientific knowledge.

The ultimate objective of this study is to enhance the existing understanding of DVT prevention, provide clinically grounded recommendations supported by evidence, and elevate the quality and safety of patient care.

DETAILED DESCRIPTION:
General Information Regarding the Thesis Topic Deep vein thrombosis (DVT) stands as a frequent complication encountered among patients undergoing on-pump cardiac surgery. A variety of interventions and protocols have been explored to forestall DVT, encompassing strategies like pharmacological prophylaxis, intermittent pneumatic leg compression, active toe movement, and supplementary measures. The objective of this survey of recent literature is to present the most current research related to nursing care protocols' impact on DVT prevention within the context of on-pump cardiac surgery patients.

Kakkos et al. (2022) undertook a thorough systematic examination, culminating in the determination that the combined utilization of intermittent pneumatic leg compression and pharmacological prophylaxis constitutes an efficacious approach for averting venous thromboembolism, encompassing DVT. Their conclusions resoundingly advocate for the integration of this dual strategy into a nursing care protocol to forestall DVT in on-pump cardiac surgery patients.

Abruzzo, Gorantla, and Thomas (2022) undertook a distinct systematic review with a focus on venous thromboembolic events in adults undergoing extracorporeal membrane oxygenation (ECMO) support. While the review did not exclusively center on on-pump cardiac surgery patients, it does offer valuable insights for managing individuals undergoing cardiac procedures. The review underlines the significance of acknowledging thromboembolic events in patients relying on ECMO support, and it underscores the importance of enacting appropriate prophylactic strategies to stave off DVT.

An, Phan, Levy, and Bruce (2016) conducted a systematic review and meta-analysis specifically focusing on hip and knee arthroplasty. Despite the different study population, their findings regarding the use of aspirin as thromboprophylaxis may have implications for on-pump cardiac surgery patients. The review emphasizes the potential of aspirin as a pharmacological intervention for preventing DVT.

In a prospective randomized study, Hickey et al. (2017) investigated the impact of active toe movement (AToM) on both calf pump function and the occurrence of DVT in patients with acute foot and ankle trauma who were treated with a cast. Although the study did not specifically target individuals undergoing on-pump cardiac surgery, it illuminates the potential advantages of integrating AToM into nursing care strategies to enhance venous return and thwart DVT. The outcomes suggest that incorporating AToM into nursing care protocols for on-pump cardiac surgery patients could hold promising benefits.

In a distinct analysis conducted by Zheng, Cheng, Wu, Wu, and Cao (2021), the authors delved into the advancements in nursing care for elderly patients who experienced postoperative hip fractures and associated DVT in China. Despite the differing study populations, this review offers insightful perspectives on nursing care protocols and optimal approaches to prevent DVT. These insights might hold relevance for on-pump cardiac surgery patients, particularly concerning nursing interventions and tactics to prevent DVT.

Ganau et al. (2017) specifically examined the risk of DVT in neurosurgery but also discussed prophylaxis protocols and best clinical practices. Although the context varies, the review emphasizes the significance of implementing appropriate prophylaxis protocols to prevent DVT. The insights from this review can be applied to on-pump cardiac surgery patients to guide nursing care protocols.

Fan et al. (2020) executed a comprehensive systematic review and meta-analysis to assess the supplementary application of intermittent pneumatic compression in hospitalized patients who were concurrently receiving pharmacologic prophylaxis for venous thromboprophylaxis. The outcomes indicate that the addition of intermittent pneumatic compression has the potential to amplify the effectiveness of pharmacologic prophylaxis. This investigation advocates for the integration of complementary interventions into nursing care protocols for the prevention of DVT in on-pump cardiac surgery patients.

In a randomized controlled trial carried out by Sakai et al. (2016), the influence of a foot pump on the incidence of DVT subsequent to total knee arthroplasty in patients undergoing treatment with edoxaban was examined. Despite the different patient demographic addressed in the study, the results underscore the prospective advantages of incorporating foot pumps as an adjunctive measure for DVT prevention. Incorporating foot pumps into nursing care protocols for on-pump cardiac surgery patients could potentially yield benefits.

Houston et al. (2020) conducted a systematic review and meta-analysis to evaluate the effectiveness and safety of tranexamic acid in high-risk non-cardiac surgical cases necessitating transfusion. Although the study's primary focus does not directly encompass on-pump cardiac surgery patients, the conclusions extend to a broader spectrum of surgical cases. The review indicates that tranexamic acid can effectively curtail bleeding and mitigate the likelihood of transfusions during high-risk surgical procedures. Considering the plausible ramifications of bleeding and subsequent immobility on DVT development, these findings may hold significance for nursing care protocols aimed at averting DVT in on-pump cardiac surgery patients.

Turan et al. (2020) executed a randomized placebo-controlled study with the intention of exploring the potential of dexmedetomidine in diminishing occurrences of atrial fibrillation and delirium subsequent to cardiac surgery. While the study focuses on distinct outcomes, it yields insights pertinent to perioperative management and interventions in cardiac surgery cases. The ramifications of atrial fibrillation and delirium on patient mobility and the risk of DVT underscore the potential value of integrating strategies to manage these complications within nursing care protocols, indirectly contributing to DVT prevention.

In their investigation, Hashemzadeh, Dehdilani, and Khanbabayi Gol (2019) delved into the impacts of basic exercise, with or without physiotherapy, in staving off DVT in postmenopausal women undergoing coronary artery bypass graft surgery. Despite the divergence in patient demographics from on-pump cardiac surgery cases, the findings underscore the significance of exercise and physiotherapy in DVT prevention. Recognizing the potential advantages of exercise and early mobilization in curtailing DVT risk, integrating these approaches into nursing care protocols for on-pump cardiac surgery patients holds potential value.

A systematic review and meta-analysis undertaken by Ho, Bham, and Pavey (2015) took a specific focus on the incidence of venous thromboembolism (VTE) and the pros and cons of thromboprophylaxis following cardiac surgery. The review furnishes invaluable perspectives regarding the overarching VTE risk and the effectiveness of thromboprophylaxis strategies. The outcomes underline the importance of well-suited thromboprophylaxis in deterring DVT in cardiac surgery patients, thereby offering informative guidance for nursing care protocols.

Shaaban and Shaaban (2021) executed a study that specifically investigated the influence of a nursing care protocol on the incidence of DVT among critically ill neurological patients. Despite the distinct patient demographic addressed, the outcomes underscore the potential advantages of nursing care protocols in mitigating DVT occurrences. The study imparts insights into the function of nursing interventions and protocols in diminishing DVT risk, which could hold relevance for on-pump cardiac surgery patients.

In an endeavor led by Sachdeva, Dalton, and Lees (2018), a systematic review and meta-analysis were conducted regarding the application of graduated compression stockings for the prevention of DVT. The review scrutinizes the efficacy of graduated compression stockings as a preventive measure. While the scope extends beyond on-pump cardiac surgery patients, the findings contribute to the comprehension of compression stockings as an intervention for DVT prevention. Incorporating the utilization of graduated compression stockings into nursing care protocols for on-pump cardiac surgery patients may offer advantages.

Khoury et al. (2020) performed a study specifically concentrating on DVT and pulmonary embolism in patients undergoing cardiac surgery. The study explores the occurrence and risk factors associated with DVT and pulmonary embolism in this specific patient population. The findings highlight the importance of identifying and addressing risk factors to prevent DVT in cardiac surgical patients, which can be valuable in shaping nursing care protocols.

Pannucci et al. (2016) conducted a systematic review that examined the pros and cons of prophylactic measures for DVT and pulmonary embolus in plastic surgery. Although the study had a different focus on a distinct surgical population, the results provide valuable insights into the potential benefits and risks linked to prophylaxis strategies. Understanding the risks associated with prophylactic measures can contribute to the development of nursing care protocols for preventing DVT in on-pump cardiac surgery patients.

Wade, Paton, and Woolacott (2016) carried out a systematic review on patient preferences and adherence to the proper usage of graduated compression stockings for DVT prevention in surgical patients. While the review does not specifically target cardiac surgery patients, it offers valuable information concerning patient preferences and adherence to compression stockings. Taking patient preferences into consideration and promoting adherence to preventive measures can enhance the effectiveness of nursing care protocols for DVT prevention.

Alaifan et al. (2019) conducted a systematic review and meta-analysis specifically focusing on tranexamic acid in cardiac surgery. Although the study focuses on a different outcome (bleeding control), it provides insights into the use of tranexamic acid, which may indirectly impact DVT prevention. Considering the potential influence of bleeding on DVT occurrence, incorporating strategies for bleeding control into nursing care protocols may indirectly contribute to DVT prevention in on-pump cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria

Patients will be eligible for participation in the study if they meet all of the following criteria:

1. Adult patients aged 18 years or older.
2. Patients scheduled to undergo elective or urgent on-pump cardiac surgery using cardiopulmonary bypass (e.g., coronary artery bypass grafting, valve replacement or repair, or combined procedures).
3. Both male and female patients.
4. Patients admitted to the participating cardiac surgery unit during the study period.
5. Patients with no evidence of preoperative deep vein thrombosis (DVT) or pulmonary embolism (PE) as confirmed by clinical assessment and/or Doppler ultrasonography when indicated.
6. Patients who are hemodynamically stable postoperatively and eligible to receive mechanical and/or pharmacological thromboprophylaxis.
7. Patients able to understand the study procedures and provide written informed consent (or consent obtained from a legal representative when applicable).
8. Patients expected to survive for at least three months postoperatively, allowing completion of the follow-up period.

Exclusion Criteria:Exclusion Criteria

Patients will be excluded from the study if they meet any of the following criteria:

1. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the previous six months.
2. Known congenital or acquired coagulation disorders, including but not limited to hemophilia, thrombophilia, or antiphospholipid syndrome.
3. Patients receiving long-term therapeutic anticoagulation (e.g., warfarin, direct oral anticoagulants) for other medical indications prior to surgery.
4. Contraindications to pharmacological thromboprophylaxis, such as:

   * Active bleeding
   * Severe thrombocytopenia (platelet count <50,000/µL)
   * History of heparin-induced thrombocytopenia (HIT)
5. Contraindications to mechanical prophylaxis, including:

   * Severe peripheral arterial disease
   * Skin ulcers, infections, or recent lower-limb surgery preventing device application
6. Patients undergoing off-pump cardiac surgery or minimally invasive cardiac procedures not requiring cardiopulmonary bypass.
7. Emergency surgery requiring immediate intervention where preoperative assessment and consent cannot be obtained.
8. Pregnant or postpartum women.
9. Patients with severe renal or hepatic failure that may interfere with anticoagulant metabolism or increase bleeding risk.
10. Patients with documented malignancy under active treatment associated with a markedly elevated thrombotic risk.
11. Patients unwilling or unable to comply with the study protocol or follow-up schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the incidence of symptomatic or confirmed deep-vein thrombosis (DVT) and/or pulmonary embolism (PE) within the 3-month follow-up period. Secondary endpoints include: adherence to the prophylaxis protocol, occurrence of prophylaxis | 3 MUNTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Facility of Nursing, Nicosia, Cyprus